CLINICAL TRIAL: NCT01781546
Title: Drug-Eluting Balloon in Stable and Unstable Angina: a Randomized Controlled Non-inferiority Trial
Brief Title: Drug-Eluting Balloon in Stable and Unstable Angina
Acronym: DEBUT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: suspeded due to slow recruitment, terminated due to interim analysis
Sponsor: North Karelia Central Hospital (Other)
Collaborators: Kuopio University Hospital (Other); University of Helsinki (Other); Turku University Hospital (Other Government); Central Hospital of Lapland, Finland (Unknown)
Responsible Party: Principal Investigator, Tuomas Rissanen, Cardiologist, MD, PhD, North Karelia Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEBUT
Record Dates: First submitted 2013-01-29; First posted 2013-02-01 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease
Keywords: drug eluting balloon; bare metal stent; coronary artery disease; acute coronary syndrome; percutaneous coronary intervention; DEB; BMS
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- drug-eluting balloon (DEB) (Experimental): Patients treated with drug-eluting balloon (DEB). Provisional stenting with BMS is permitted in case of a flow-limiting dissection or significant recoil (>30% in main branch and >50% side-branch), Includes both stable CAD and ACS patients.
  Interventions: Procedure: drug-eluting balloon (DEB)
- bare-metal stent (BMS) (Active Comparator): Patients treated with bare-metal stent (BMS). Includes both stable CAD and ACS patients.
  Interventions: Procedure: bare-metal stent (BMS)

INTERVENTIONS:
Procedure: drug-eluting balloon (DEB) — The length of the DEB is chosen so that the lesion and 2mm from both ends are covered by the DEB. If needed, several DEBs can be used to cover the whole lesion. The diameter of the DEB and the pressure used is chosen so that the balloon-artery -ratio is 0.8-1.0. In case of a flow limiting dissection, significant recoil or coronary perforation, a provisional BMS is implanted (stent-artery -ratio 1.1) and the post dilatation is performed if indicated (the lesion length is >20mm or stent malapposition is suspected).
  Other Names: SeQuent Please (B Braun, Germany, diameter 2,5-4.0mm)
  Arms: drug-eluting balloon (DEB)
Procedure: bare-metal stent (BMS) — The BMS is implanted after predilatation (stent-artery -ratio 1.1) to cover the whole lesion and the postdilatation is performed if indicated (the lesion length >20mm or stent malapposition is suspected).
  Other Names: Integrity stent (Medtronic, USA, diameter 2,5-4,0mm)
  Arms: bare-metal stent (BMS)

SUMMARY:
The purpose of this study is to compare DEB with BMS in CAD patients who are at high risk of bleeding and in whom the use of DES is therefore avoided. Our hypothesis is that PCI with DEB is non-inferior to BMS in the treatment of stable CAD or in ACS (UAP or NSTEMI) in patients at high risk of bleeding.

DETAILED DESCRIPTION:
Stenting has reduced the need of revascularization procedures in stable CAD and ACS as compared to POBA. The use of stents is favored in stable CAD and in ACS according the the present ESC guidelines. However, especially in patients on warfarin or in patients at a high bleeding risk, stenting (and the use of DES in particular) is not recommended because of the longer DAPT required. In these patients, BMS may be used to shorten the duration of DAPT. However, there are problems associated with the treatment using BMS. First of all, a considerable high rate of restenosis is associated with stenting with BMS. Furthermore, stenting may be complicated by the "no-reflow" phenomenon, a coronary dissection or the closure of side branch during the treatment of bifurcation lesions. Implantation of a stent also exposes the patient to stent thrombosis. In contrast, these problems may be avoided by the use of DEB with the provisional BMS strategy.

The use of DEB has already been established in the treatment of ISR. Despite the lack of data of RCTs, DEB is already widely used in a variety of clinical situations in which stenting is not desirable. These situations include for example anticoagulation treatment, a high bleeding risk, poor compliance regarding medication, small vessels, bifurcation lesions, long and/or calcified lesions, in case of a marked variation in the vessel reference caliber, in long lesions and in patients with ACS. The all-comer registry data is promising but only hypothesis generating. Thus, it would be very important and ethical to test the efficacy of DEB in a wider patient population in a randomized controlled study.

Our hypothesis is that DEB is non-inferior to BMS in the treatment of stable CAD or in ACS (UAP or NSTEMI) in patients on anticoagulation medication or otherwise having a high bleeding risk. Our study sheds light on the use of DEB in PCI of this challenging patient population. In most previous studies, BMS has been routinely added to the DEB treatment. This strategy seems not to yield any benefit but in contrast causes an increased risk of restenosis as compared to the DEB only strategy with provisional stenting. Finally, the current data on the use of DEB in patients with ACS is scarce and our study gives significant information also on this important issue.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed written consent
* At least one of the following

  1. Patient is using oral anticoagulation (warfarin, dabigatran or rivaroxaban)
  2. Anemia (hemoglobin below the threshold: < 117g/l in women and < 134 g/l in men) or thrombocytopenia (<100) detected <6 months prior the PCI
  3. Active malign disease (metastatic cancer or ongoing radio- or chemotherapy)
  4. Prior intracerebral hemorrhage or ischemic stroke
  5. Severe kidney or liver dysfunction (eGFR < 30ml/kg/min, liver cirrhosis, BIL >2x over threshold or ALAT >3x over threshold)
  6. Elective surgery planned < 12 months after the PCI
  7. General frailty for e.g. because of long corticosteroid treatment or generalized cachexia (BMI < 20 kg/m2)
  8. Age ≥ 80 years
  9. Inability or suspected inability to use DAPT for 12 months
* Either of the following:

  10) Prior bleeding (BARC 2-5)
  1. Stable angina or dyspnea and a coronary narrowing causing myocardial ischemia detected in the angiogram. Ischemia is documented by the pressure wire measurement (FFR) or by a non-invasive test such as stress ECG test or perfusion imaging
  2. ACS (UAP or NSTEMI): symptoms of heart ischemia ≥ 20 minutes and ≥ 0,5mm ST-depression or transient ST-elevation or T-wave inversion at least in two adjacent leads and/or a high sensitivity troponin (hs-tnt) rise at least one unit above the 99. percentile or at least 50% rise in hs-tnt between two samples taken 3 hours apart
* ≥1 de novo lesions in native coronary arteries or bypass vein grafts
* Reference diameter of the vessel is 2,5-4,0mm
* Lesion or lesions are suitable for PCI

Exclusion Criteria:

* Inability to give written consent
* STEMI
* Reference diameter of the vessel is <2,5mm or >4,0mm
* Bifurcation lesion requiring the stenting of the side branch
* Dissection affecting the flow (TIMI<3) or significant recoil (>30% in main branch, >50% in side branch) after predilatation
* In-stent restenosis
* Life expectancy < 12 months
* Cardiogenic shock at the arrival to the coronary angiography
* Uncertainty about neurological recovery e.g. after resuscitation
* Unprotected left main (LM) lesion
* Chronic total occlusion (CTO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-05-22 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
MACE (Major Adverse Cardiac Event = a composite of cardiac death, nonfatal myocardial infarction (MI) and ischemia driven target lesion revascularization (ID-TLR)) | At 9 months
  In stable patients, the evidence of ischemia is acquired either by non-invasive testing (for example stress ECG or perfusion imaging) or by pressure wire measurement (FFR) during coronary angiography.
ID-TLR (Ischemia Driven Target Lesion Revascularisation) | at 36 months

SECONDARY OUTCOMES:
ID-TLR (Ischemia Driven Target Lesion Revascularisation) | At 9 months
Failure to treat the lesion | During PCI
  The failure to deliver the randomized treatment (DEB or BMS) to the target lesion is defined as a failure to treat the lesion.

OTHER OUTCOMES:
Control angiography and OCT imaging | At 6 months
  30 patients (15 from each group) will be randomly invited to a control angiography and OCT imaging to asses the rate of restenosis and endothelial healing.
MACE (Major Adverse Cardiac Event = a composite of cardiac death, nonfatal myocardial infarction (MI) and ischemia driven target lesion revascularization (ID-TLR)) | at 36 months
ID-TLR (Ischemia Driven Target Lesion Revascularisation) | at 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Rissanen, MD, PhD, Principal Investigator — North Karelia Central Hospital; Antti Siljander, MD, Principal Investigator — North Karelia Central Hospital
Locations (4):
- Finland (4):
  - Helsinki University Hospital Heart Center, Helsinki
  - North Karelia Central Hospital, Joensuu
  - Kuopio University Hospital, Kuopio
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Rissanen TT, Uskela S, Eranen J, Mantyla P, Olli A, Romppanen H, Siljander A, Pietila M, Minkkinen MJ, Tervo J, Karkkainen JM; DEBUT trial investigators. Drug-coated balloon for treatment of de-novo coronary artery lesions in patients with high bleeding risk (DEBUT): a single-blind, randomised, non-inferiority trial. Lancet. 2019 Jul 20;394(10194):230-239. doi: 10.1016/S0140-6736(19)31126-2. Epub 2019 Jun 13. PMID 31204115